CLINICAL TRIAL: NCT04601519
Title: Effect of Type 1 Diabetes on Sleep Fragmentation
Acronym: DIAPASOM5
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC18.271; 2018-A02474-51 (Other: ID RCB)
Record Dates: First submitted 2020-10-16; First posted 2020-10-23 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2020-10

CONDITIONS: Type 1 Diabetes
Keywords: Type1 diabetes; Sleep fragmentation and quality of sleep; the nocturia; the hypoglycemias; the hyperglycemias
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Sleep Deprivation; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients-type 1 diabetes: Participants are recruited by e-mail, among the users of the libreview platform (Abbott), who are followed up for type 1 diabetes at the CHU Grenoble Alpes (France), to participate in an anonymous online questionnaire and to allow their glycemic data extracted from the libreview platform to be used for the research.
  Interventions: Other: Cross-sectional observational study

INTERVENTIONS:
Other: Cross-sectional observational study — Online questionnaire on the impact of type 1 diabetes on sleep quality
  Other Names: Online questionnaire

SUMMARY:
The main objective of this study is the objective evaluation of disease related sleep fragmentation in subjects with type 1 diabetes.

DETAILED DESCRIPTION:
The influence of sleep duration and sleep schedules (social jetlag) on glycemic control in type 1 diabetes has been shown in several previous studies, including by the investigators of this study.

Following these publications, patients have expressed the opinion via social networks that type 1 diabetes disease is itself a factor that alters the quality of sleep. Indeed, it appears that the cross-sectional studies published to date have focused on the association between the subjects' sleep habits and the balance of their diabetes, without having questioned the role of the pathology on sleep quality.

The main objective of this study is the objective evaluation of disease related sleep fragmentation in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported type 1 diabetes
* Male or female
* Self-reported age > 18 years old
* Subject user of a freestyle capillary meter

Exclusion Criteria:

* Opposition to Use of Data for Teaching and Research Purposes
* Other type of diabetes
* Self-reported age under 18 years of age
* Subject non-user of a freestyle capillary meter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients having a self-reported type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective sleep fragmentation | 1 week
  Number of nocturnal awakenings objectively measured by the number of voluntary glycemia tests performed during the sleep period, according to freestyle recordings.

SECONDARY OUTCOMES:
Subjective sleep fragmentation | 1week
  Number of self-reported awakenings by patients
Subjective sleep quality | 1 week
  Analogical scale (from 0 to 10) to grade overall sleep quality
Subjective impact of type 1 diabetes on sleep quality. | 1 week
  Analogical scale (from 0 to 10) to grade overall sleep quality
Sleep fragmentation by subgroups | 1 week
  Comparison of the number of nocturnal awakenings due to the disease between the following subgroups :
  * Men versus women
  * By age categories (quartiles)
  * According to diabetes control

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure Borel, MD, PhD, Principal Investigator — Grenoble Alpes university hospital
Locations (1):
- Grenoble Alpes university hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided
There is a plan to make IPD and related data dictionaries available to perform meta-analyses based on individual data.
  The sharing of data will need the acceptation by the Principal Investigator.

REFERENCES:
- [Background] Larcher S, Gauchez AS, Lablanche S, Pepin JL, Benhamou PY, Borel AL. Impact of sleep behavior on glycemic control in type 1 diabetes: the role of social jetlag. Eur J Endocrinol. 2016 Nov;175(5):411-9. doi: 10.1530/EJE-16-0188. Epub 2016 Aug 16. PMID 27530460
- [Background] Larcher S, Benhamou PY, Pepin JL, Borel AL. Sleep habits and diabetes. Diabetes Metab. 2015 Sep;41(4):263-271. doi: 10.1016/j.diabet.2014.12.004. Epub 2015 Jan 23. PMID 25623152
- [Background] Borel AL, Pepin JL, Nasse L, Baguet JP, Netter S, Benhamou PY. Short sleep duration measured by wrist actimetry is associated with deteriorated glycemic control in type 1 diabetes. Diabetes Care. 2013 Oct;36(10):2902-8. doi: 10.2337/dc12-2038. Epub 2013 May 28. PMID 23715755
- [Background] Borel AL, Benhamou PY, Baguet JP, Debaty I, Levy P, Pepin JL, Mallion JM. Short sleep duration is associated with a blood pressure nondipping pattern in type 1 diabetes: the DIAPASOM study. Diabetes Care. 2009 Sep;32(9):1713-5. doi: 10.2337/dc09-0422. Epub 2009 Jun 19. PMID 19542208